CLINICAL TRIAL: NCT06347926
Title: Study of Sexual Quality of Life in Women With Breast Cancer Who Had Multidisciplinary Management With Photobiomodulation for Genitourinary Syndrome of the Menopause
Acronym: EVABIOSEIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut du Cancer de Montpellier - Val d'Aurelle (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PROICM 2023-11 EVA
Record Dates: First submitted 2024-03-28; First posted 2024-04-04 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: Sexual troubles; Irritation; Dyspareunia; Vaginal dryness; Photobiomodulation
MeSH Terms: conditions — Breast Neoplasms; Dyspareunia

STUDY DESIGN:
Intervention Model Description: Questionnaires given before and after photobiomodulation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Questionnaires, scale and score (Experimental): Questionnaires, numeric visual scale and clinical score
  Interventions: Procedure: Questionnaires given before and after photobiomodulation

INTERVENTIONS:
Procedure: Questionnaires given before and after photobiomodulation — Questionnaires given at 1 month, 6 months and 12 months

SUMMARY:
The treatment of breast cancer as well as the disease are responsible for genito-urinary symptoms that can persist over time and impair quality of life. Given the improved prognosis of breast cancer, more and more patients are confronted with specific post-cancer issues, and the care has become a major health challenge.

Sexual health is a crucial component of well-being and overall quality of life. Vaginal dryness and dyspareunia are symptoms frequently found in patients treated for breast cancer, with chemotherapy and hormone therapy as risk factors. However, the treatment of sexual disorders remains underdeveloped in France.

Vaginal dryness is part of a broader syndrome known as genitourinary syndrome of menopause (GSM), or vulvovaginal atrophy, which may combine vulvovaginal (dryness, irritation, burning), sexual (dyspareunia) and urinary (infections, pollakiuria, urgency) symptoms secondary to hypoestrogenemia, exacerbated by breast cancer treatments. Since hormonal treatments are contraindicated, the first-line treatment for GSM in patients treated for breast cancer is the application of non-hormonal trophic treatments (regular vaginal moisturizers, lubricants during intercourse). However, these treatments are often insufficient to provide effective relief. There is therefore growing interest in the development of second-line treatments for GSM : intra-vaginal hyaluronic acid injections, laser, photobiomodulation (PBM), etc. PBM using Light Emitting Diodes (LED) has been proposed as an alternative treatment for genitourinary syndrome of the menopause. The tissues are exposed to light sources in the visible spectrum, inducing non-thermal, non-cytotoxic biological effects that improve vaginal tissue trophicity.

In line with previous studies of sexual quality of life carried out at the center, and in the context of the recent establishment of our multidisciplinary network for the 2nd-line treatment of genitourinary menopausal syndrome with Photobiomodulation, we would like to carry out a descriptive study of the sexual QoL of patients undergoing treatment for breast cancer and benefiting from this oncosexological support.

DETAILED DESCRIPTION:
Breast cancer affects around one in eight women, accounting for 58,459 new cases in 2018 in France. Advances in treatment have improved overall survival, which is currently around 90% at 5 years in industrialized countries. In France, 5.3% of women have survived breast cancer.

However, the disease and its treatment are responsible for symptoms that can persist over time and impair quality of life. Given the improved prognosis of breast cancer, more and more patients are confronted with the specific problems of the post-cancer period, and care for them has become a major health issue, highlighted in international recommendations and in Cancer Plans since 2003.

Sexual health is a crucial component of well-being and overall quality of life. Sexual quality of life is frequently impaired after cancer treatment. A large-scale survey carried out in France showed that sexual quality of life remained impaired in almost two thirds of patients 2 years and 5 years after cancer diagnosis, all sites combined. An abundance of literature underlines the high frequency of sexuality and intimacy disorders in patients treated for breast cancer, from diagnosis, throughout treatment and into the post-cancer period.

Sexual health is a complex issue, influenced by multiple factors such as education, beliefs, socio-cultural factors, intimacy, relationship with partner, physical and psychological well-being, body image, and personal and gender identity. These multiple factors can be disrupted, modified and altered as a result of cancer diagnosis and treatment. Vaginal dryness and dyspareunia are symptoms frequently found in patients treated for breast cancer, with chemotherapy and hormone therapy as risk factors.

However, the management of sexual disorders remains underdeveloped in France. Three prospective studies have been carried out at the Institute of Cancer in Montpellier (ICM), two of which have been published, analyzing sexual quality of life in patients with non-metastatic breast cancer, and have shown a deterioration in sexual quality of life similar to that described in the literature, with in particular a high frequency of libido disorders, vaginal dryness and altered sexual satisfaction. A low level of communication between patients and healthcare professionals was reported, with a high demand for care expressed by patients. Patients' opinions and suggestions for optimal care were also collected and analyzed. The analysis of these data showed that patients had initiated first-line treatments for vaginal dryness.

Vaginal dryness is part of a broader syndrome known as genitourinary syndrome of menopause (GSM), or vulvovaginal atrophy, which may combine vulvovaginal (dryness, irritation, burning), sexual (dyspareunia) and urinary (infections, pollakiuria, urgency) symptoms secondary to hypoestrogenemia, exacerbated by breast cancer treatments. Since hormonal treatments are contraindicated, the first-line treatment for GSM in patients treated for breast cancer is the application of non-hormonal trophic treatments (regular vaginal moisturizers, lubricants during intercourse). However, these treatments are often insufficient to provide effective relief. There is therefore growing interest in the development of second-line treatments for GSM : intra-vaginal hyaluronic acid injections, laser, photobiomodulation (PBM), etc. Light Emitting Diode (LED) PBM has been proposed as an alternative treatment for genitourinary menopausal syndrome. he tissues are exposed to light sources in the visible spectrum, inducing non-thermal, non-cytotoxic biological effects that improve vaginal tissue trophicity. This non-invasive technique has few contraindications (epilepsy, photosensitizing treatment) and no known serious side effects, and has been studied in a number of indications, notably for the treatment of oral mucositis. There are few data on vaginal application, and this technology is being evaluated as part of a clinical trial at the Nimes hospital in patients with GSM in the general population. Interim results based on the inclusion of 130 patients showed clinical improvement in 61 out of 100 patients ("better" or "much better") treated with 6 sessions of PBM, with no serious adverse effects (PhD thesis). There are currently no data specifically on women treated for breast cancer. In the context of setting up an oncosexology care network at the Institute of Cancer in Montpellier.

In line with previous studies of sexual QoL carried out at the center, and in the context of the recent establishment of our multidisciplinary network for the 2nd-line treatment of genitourinary menopausal syndrome with Photobiomodulation, we would like to carry out a descriptive study of the sexual Qaulity of life of patients undergoing treatment for breast cancer and benefiting from this oncosexological support.

ELIGIBILITY:
Inclusion Criteria:

1. Woman ≥ 18,
2. Diagnosis of breast cancer regardless of tumor biology or stage (localized or metastatic),
3. Patient with persistent menopause genito-urinary symptoms after a minimum of 3 months of local treatment with vaginal moisturizers,
4. Patient eligible for photobiomodulation as 2nd-line treatment for menopausal genitourinary syndrome as part of routine care.

Exclusion Criteria:

1. Patient who have already undergone or are undergoing a 2nd-line treatment for menopause genito-urinary symptoms (photobiomodulation, laser, intra-vaginal injection of hyaluronic acid, etc.),
2. Patient with psychic or cognitive impairment, or not sufficiently fluent in French to be able to fill in the quality of life questionnaires.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Sexual satisfaction score on one dimension of the SHQ-22 questionnaire | From baseline to 1 year
  Evaluation by sexual health questionnaire (SHQ-22). The SHQ-22 questionnaire is a multidimensional quality of life instrument used to measure sexual health in patients with cancer (men or women). This new tool covers both sexual functioning and psychosexual components. It includes 8 items on sexual satisfaction, 3 items on sexual pain, and 11 single items in an integrative approach, leading to 7 functional scales and 4 symptom scales. In these questionnaires, higher scores in the functioning scales indicate a better functional level, whereas higher scores in the symptom scales indicate the severity of problems.

SECONDARY OUTCOMES:
Sexual quality of life scores obtained on all dimensions of the SHQ-22 questionnaire | From baseline to 1 year
  Evaluation by sexual health questionnaire (SHQ-22). The SHQ-22 questionnaire is a multidimensional quality of life instrument used to measure sexual health in patients with cancer (men or women). This new tool covers both sexual functioning and psychosexual components. It includes 8 items on sexual satisfaction, 3 items on sexual pain, and 11 single items in an integrative approach, leading to 7 functional scales and 4 symptom scales. In these questionnaires, higher scores in the functioning scales indicate a better functional level, whereas higher scores in the symptom scales indicate the severity of problems.
Patient Global Impression of Improvement (PGI-I) score | From baseline to 1 year
  Evaluation by questionnaire Patient Global Impression of Improvement (PGI-I). The PGI-I is a transition scale that is a single question asking the patient to rate their urinary tract condition now, as compared with how it was prior to before beginning treatment on a scale from 1 to 7. Very much better (1) to Very much worse (7).
Determination of the Vaginal Health Index clinical score | From baseline to 1 year
  The vaginal health index scores five different signs of vaginal health on a one-to-five ranking system. The lower your score, the more unhealthy your vaginal tissue is. The score ranges from 5 (the worst vaginal health) to 25 (the best vaginal health). This scoring system helps doctors to diagnose the severity of genitourinary syndrome of menopause.
Determination of symptoms of vulvovaginal atrophy by a visual numerical scale | From baseline to 1 year
  Visual numerical scale from 0 (no pain and discomfort) to 10 (the most intense pain and discomfort)
Determination of adverse events by using Common Terminology Criteria for Adverse Events (CTCAE) scale of the National Cancer Institute. | From baseline to 1 year
Number of patients taking other treatments for treating sexual troubles | From baseline to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Angélique Bobrie, MD, Study Chair — Institute of Cancer in Montpellier
Locations (1):
- Institute of Cancer in Montpellier, Montpellier, Hérault, France

IPD SHARING:
Plan to Share IPD: Yes
Participant data will be made available on request and with the completion of a contract between the sponsor and the requester.
Supporting Information: Study Protocol
Time Frame: Access to study data upon written detailed request sent to the institute of Montpellier Cancer (ICM), following publication and until 5 years after publication of summary data.
Access Criteria: The data shared will be limited to that required for independent mandated verification of the published results, the applicant will need authorization from ICM for personal access, and data will only be transferred after signing of a data access agreement.

REFERENCES:
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Allemani C, Matsuda T, Di Carlo V, Harewood R, Matz M, Niksic M, Bonaventure A, Valkov M, Johnson CJ, Esteve J, Ogunbiyi OJ, Azevedo E Silva G, Chen WQ, Eser S, Engholm G, Stiller CA, Monnereau A, Woods RR, Visser O, Lim GH, Aitken J, Weir HK, Coleman MP; CONCORD Working Group. Global surveillance of trends in cancer survival 2000-14 (CONCORD-3): analysis of individual records for 37 513 025 patients diagnosed with one of 18 cancers from 322 population-based registries in 71 countries. Lancet. 2018 Mar 17;391(10125):1023-1075. doi: 10.1016/S0140-6736(17)33326-3. Epub 2018 Jan 31. PMID 29395269
- [Background] Carter J, Lacchetti C, Andersen BL, Barton DL, Bolte S, Damast S, Diefenbach MA, DuHamel K, Florendo J, Ganz PA, Goldfarb S, Hallmeyer S, Kushner DM, Rowland JH. Interventions to Address Sexual Problems in People With Cancer: American Society of Clinical Oncology Clinical Practice Guideline Adaptation of Cancer Care Ontario Guideline. J Clin Oncol. 2018 Feb 10;36(5):492-511. doi: 10.1200/JCO.2017.75.8995. Epub 2017 Dec 11. PMID 29227723
- [Background] Ben Charif A, Bouhnik AD, Courbiere B, Rey D, Preau M, Bendiane MK, Peretti-Watel P, Mancini J. Sexual health problems in French cancer survivors 2 years after diagnosis-the national VICAN survey. J Cancer Surviv. 2016 Jun;10(3):600-9. doi: 10.1007/s11764-015-0506-3. Epub 2015 Dec 21. PMID 26685697
- [Background] Seguin L, Touzani R, Bouhnik AD, Charif AB, Marino P, Bendiane MK, Goncalves A, Gravis G, Mancini J. Deterioration of Sexual Health in Cancer Survivors Five Years after Diagnosis: Data from the French National Prospective VICAN Survey. Cancers (Basel). 2020 Nov 20;12(11):3453. doi: 10.3390/cancers12113453. PMID 33233583
- [Background] Dizon DS. Quality of life after breast cancer: survivorship and sexuality. Breast J. 2009 Sep-Oct;15(5):500-4. doi: 10.1111/j.1524-4741.2009.00766.x. Epub 2009 Jul 14. PMID 19614908
- [Background] Frechette D, Paquet L, Verma S, Clemons M, Wheatley-Price P, Gertler SZ, Song X, Graham N, Dent S. The impact of endocrine therapy on sexual dysfunction in postmenopausal women with early stage breast cancer: encouraging results from a prospective study. Breast Cancer Res Treat. 2013 Aug;141(1):111-7. doi: 10.1007/s10549-013-2659-y. Epub 2013 Aug 14. PMID 23942873
- [Background] Del Pup L, Villa P, Amar ID, Bottoni C, Scambia G. Approach to sexual dysfunction in women with cancer. Int J Gynecol Cancer. 2019 Mar;29(3):630-634. doi: 10.1136/ijgc-2018-000096. Epub 2019 Feb 13. PMID 30765487
- [Background] Ribi K, Luo W, Bernhard J, Francis PA, Burstein HJ, Ciruelos E, Bellet M, Pavesi L, Lluch A, Visini M, Parmar V, Tondini C, Kerbrat P, Perello A, Neven P, Torres R, Lombardi D, Puglisi F, Karlsson P, Ruhstaller T, Colleoni M, Coates AS, Goldhirsch A, Price KN, Gelber RD, Regan MM, Fleming GF. Adjuvant Tamoxifen Plus Ovarian Function Suppression Versus Tamoxifen Alone in Premenopausal Women With Early Breast Cancer: Patient-Reported Outcomes in the Suppression of Ovarian Function Trial. J Clin Oncol. 2016 May 10;34(14):1601-10. doi: 10.1200/JCO.2015.64.8675. Epub 2016 Mar 28. PMID 27022111
- [Background] Aptecar L, Fiteni F, Jarlier M, Delaine S, Guillerme V, Jacot W, D'Hondt V. Prospective evaluation of sexual health in breast cancer women during the first year of adjuvant hormonal treatment using a cancer patient's dedicated questionnaire: A glaring gap of communication between health professionals and patients. Breast Cancer Res Treat. 2021 Apr;186(3):705-713. doi: 10.1007/s10549-020-06062-x. Epub 2021 Jan 15. PMID 33452553
- [Background] Bobrie A, Jarlier M, Moussion A, Jacot W, D'Hondt V. Sexual quality of life assessment in young women with breast cancer during adjuvant endocrine therapy and patient-reported supportive measures. Support Care Cancer. 2022 Apr;30(4):3633-3641. doi: 10.1007/s00520-022-06810-3. Epub 2022 Jan 14. PMID 35028721
- [Background] Hocke C, Diaz M, Bernard V, Frantz S, Lambert M, Mathieu C, Grellety-Cherbero M. [Genitourinary menopause syndrome. Postmenopausal women management: CNGOF and GEMVi clinical practice guidelines]. Gynecol Obstet Fertil Senol. 2021 May;49(5):394-413. doi: 10.1016/j.gofs.2021.03.025. Epub 2021 Mar 20. French. PMID 33757926
- [Background] Maris E, Salerno J, Hedon B, Mares P. [Management of vulvovaginal atrophy: Physical therapies. Postmenopausal women management: CNGOF and GEMVi clinical practice guidelines]. Gynecol Obstet Fertil Senol. 2021 May;49(5):414-419. doi: 10.1016/j.gofs.2021.03.021. Epub 2021 Mar 20. French. PMID 33757917
- [Background] Lanzafame RJ, de la Torre S, Leibaschoff GH. The Rationale for Photobiomodulation Therapy of Vaginal Tissue for Treatment of Genitourinary Syndrome of Menopause: An Analysis of Its Mechanism of Action, and Current Clinical Outcomes. Photobiomodul Photomed Laser Surg. 2019 Jul;37(7):395-407. doi: 10.1089/photob.2019.4618. Epub 2019 Jun 17. PMID 31210575